CLINICAL TRIAL: NCT01766596
Title: Study the Signs of Ocular Degeneration in a Population Cohort (Dijon 3C Montrachet Cohort): Seek Correlations Between Signs of Neurological and Vascular Degeneration and Signs of Ocular Aging
Brief Title: Study the Signs of Ocular Degeneration in a Population Cohort (Dijon 3C Montrachet Cohort)
Acronym: 3C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Creuzot-Garcher PHRC IR 2009
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: AMD; Glaucoma
Keywords: Ophthalmology; Age-related ocular pathologies
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

ARMS (1):
- 3C cohort (Other)
  Interventions: Procedure: Optical Coherence Tomography

INTERVENTIONS:
Procedure: Optical Coherence Tomography

SUMMARY:
The aim of the study proposed in Dijon is above all to focus on the possible relationship between age-related ocular pathologies (AMD and glaucoma) and et les degenerative neurological and cardiac pathologies.

The principal objective is to seek in subjects who have undergone cerebral MRI and echocardiography, associations between the thickness of postganglionic fibers measured by Optical Coherence Tomography at the 7th year (n=1500) and signs of cerebral impairment (psycho-cognitive tests, circulation time, MRI signs). This association will be studied after taking into account the principal environmental (particularly dietary) and genetic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have given their written consent
* Persons who are taking part in the Dijon 3C study

Exclusion Criteria:

* Persons who are not registered with social security agency
* Persons who are unable to sit upright during a consultation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Measure the mean thickness of postganglionic fibers | T=7 years of the 3C cohort
  Measure the thickness of postganglionic fibers by Optical Coherence Tomography in the 4 quadrants of the peripapillary sclera.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France